CLINICAL TRIAL: NCT03958461
Title: Connection Between Periodontitis and Exudative Age-related Macular Degeneration
Acronym: FLAREPARO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Petteri Karesvuo, Principal Investigator, M.D. FEBO, Specialist in Ophthalmology, University of Helsinki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRRG FLAREPARO
Record Dates: First submitted 2019-05-15; First posted 2019-05-22 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Periodontitis
Keywords: periodontitis; exudative age-related macular degeneration; wet age-related macular degeneration; AMD; BAB; aqueous flare
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Calculus removement (Other): Anti-infective treatment of teeth
  Interventions: Procedure: Anti-infective treatment of periodontal pockets

INTERVENTIONS:
Procedure: Anti-infective treatment of periodontal pockets — Removing calculi from teeths' periodontal pockets

SUMMARY:
Aqueous flare is increased in different kind of inflammations of eye. This is caused by disruption of blood-aqueous-barrier. The investigators assume that low grade systemic inflammation, such as periodontitis, increase aqueous flare and possibly activates exudative age-related macular degeneration.

DETAILED DESCRIPTION:
Periodontitis is a chronic low-grade bacterial infection of supporting tissue of teeth. Chronic periodontitis is often non symptomatic. Inflammation is located usually in deepened periodontal pockets (> 4mm or >6mm) and it leads to alveolar bone loss and eventually detachment of teeth. In Finland, it is estimated that 64% of people have mild form of periodontitis and severe form approximately 21% according to Health 2000 and Health 2011 studies. Various gram negative and positive pathogens have been isolated in infected area, Porhyromonas Gingivalis, Prevotella intermedia, Treponema denticola, Tannerella forsynthesis, Campylobacter rectus, Aggregatibacter actinomycetemcomitans and Peptostreoptococcus micros. Periodontitis causes endotoxemia in circulation via inflamed supporting structure of teeth. Endotoxins such as lipopolysaccharide (LPS) and their concentrations are elevated in blood and it is found that C-reactive protein (CRP), interleukins and cytokines are also elevated in blood due to periodontitis. As a result periodontitis activates low-grade systemic inflammation and complement system activation classical and alternative pathway. In some studies, the treatment of periodontitis diminished CRP values and lowered the systemic inflammation. Periodontitis has been connected with many diseases, such as atherosclerosis, coronary artery disease, Alzheimer's disease and adverse pregnancy outcomes. Furthermore, various studies have found association between periodontitis and age-related macular degeneration. Severity of diabetic retinopathy was linked with severity of periodontitis furthermore scleritis was resoluted after periodontal treatment Aqueous flare is a hallmark of blood-aqueous-barrier. Increased aqueous flare is found in different types of inflammations and infections of eye for example in iritis and in endophthalmitis. In addition intraocular surgery promotes almost always aqueous flare postoperatively. Increased aqueous flare and macular thickening and postoperative cystoid macular edema (PCME) are found after uneventful cataract operation. The higher flare levels correlated with the activity in wet age-related macular degeneration and in addition in central retinal vein occlusion.

Here in this study the investigators aimed to characterize the association between the periodontitis and elevated aqueous flare values as a potential risk factor for developing exudative macular degeneration.

Material and methods Study will be conducted at Kymenlaakso Central Hospital in Kotka, Finland. Time period is going to be between 1.6.2019-1.6.2021. One hundred participents will be enrolled in this study calculated with power analysis (0.8). Drop-out patients will be about 5%. The investigators will measure periodontal pockets (>4mm or >6mm) and number of affected teeth and give anti-infective treatment in addition to taking bacterial PCR samples. Follow up visits will be after 6 weeks.

Non-invasive and safe aqueous flare measurements will be performed by investigators with aqueous flare meter (FM-600 Kowa Company, Ltd., Nagoya, Japan) before and 1 hour after anti-infective treatment. The flare values varies between < 10 photon units pu/msec in healthy subjects without BAB disruption and over 300 pu/msec in eyes with severe BAB disruption. Automated reliability analysis of the measurements performed by the laser flare meter will be taken into account. The patient information will be stored in a password protected computer and no one else outside the study is not allowed to participate the study and process the data. Study material will be processed in a HUS computer or in a password protected personal computer via VPN communication link. Helsinki University Helpdesk will offer user interface. Participents personal infromation will be deleted after usage and anonymous registry and data will be stored for 5 years in a digital password protected SSD memory after the publication of the study findings.

Ethical perspectives The treatment models used in the study comply with Good Clinical Practice. The patient will be provided with both verbal and written information before signing the consent form. Study subjects may withdraw their consent after the study has begun. The study will have no effect in any way on the care that the patient receives. Information about the study subject and the results obtained from the study will be handled confidentially. The study aims to provide the latest definitive results, nor can it be conducted in any other way. The study may have a significant benefit on understanding wet AMD pathophysiology. The study will follow the principles of the Declaration of Helsinki of the World Medical Association.

ELIGIBILITY:
Inclusion Criteria:

* periodontitis

Exclusion Criteria:

* no periodontitis, any eye disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
<10pu/msec to over 300pu/msec | Change from Baseline aqueous flare value at 6 weeks
  Aqueous flare value before (in the same day) and after 6 weeks of anti-infective treatment of teeth

CONTACTS AND LOCATIONS:
Overall Officials: Raimo Tuuminen, PhD, Study Chair — Helsinki Retina Research Group; Minna Karesvuo, DDS, Study Director — University of Helsinki
Locations (1):
- Kymeenlaakson keskussairaala, Kotka, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shin YU, Lim HW, Hong EH, Kang MH, Seong M, Nam E, Cho H. The association between periodontal disease and age-related macular degeneration in the Korea National health and nutrition examination survey: A cross-sectional observational study. Medicine (Baltimore). 2017 Apr;96(14):e6418. doi: 10.1097/MD.0000000000006418. PMID 28383406
- [Background] Wagley S, Marra KV, Salhi RA, Gautam S, Campo R, Veale P, Veale J, Arroyo JG. PERIODONTAL DISEASE AND AGE-RELATED MACULAR DEGENERATION: Results From the National Health and Nutrition Examination Survey III. Retina. 2015 May;35(5):982-8. doi: 10.1097/IAE.0000000000000427. PMID 25627087
- [Background] Karesvuo P, Gursoy UK, Pussinen PJ, Suominen AL, Huumonen S, Vesti E, Kononen E. Alveolar bone loss associated with age-related macular degeneration in males. J Periodontol. 2013 Jan;84(1):58-67. doi: 10.1902/jop.2012.110643. Epub 2012 Mar 13. PMID 22414258